CLINICAL TRIAL: NCT03341936
Title: Neodjuvant Nivolumab and Lirilumab, Followed by Surgery, Followed by Adjuvant Nivolumab and Lirilumab, in Patients With Relapsed, Resectable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Neodjuvant Nivolumab and Lirilumab, Followed by Surgery, Followed by Adjuvant Nivolumab and Lirilumab, in SCCHN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-411
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Results first posted 2022-06-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Nivolumab; lirilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Lirilumab (Experimental): * The drugs will be administered intravenously. A single dose of Nivolumab and Lirilumab will be administered prior Salvage surgical resection.
  * In Cycle 1-3: Nivolumab will be administered on Days 1 and 15 and lirilumab will be administered on Day 1 of each 28 day long cycle
  * In Cycle 4-6 and beyond: Nivolumab and lirilumab will be administered on Day 1 of each 28 day long cycle.
  Interventions: Drug: Nivolumab; Drug: Lirilumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells
Drug: Lirilumab — Lirilumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells

SUMMARY:
This research study is studying a combination of two immunotherapy drugs, as a possible treatment for locoregionally recurrent squamous cell carcinoma of the head and neck.

The immunotherapy drugs involved in this study are:

* Nivolumab (Opdivo™)
* Lirilumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or combination of drugs to learn whether it works in treating a specific disease. "Investigational" means that the drug/s is being studied.

The purpose of this study is to evaluate effectiveness (how well the drug/s work) of nivolumab in combination with lirilumab in participants with SCCHN.

Nivolumab and lirilumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells. Both nivolumab and lirilumab have been demonstrated to activate the immune system to attack cancer cells in participants with different types of cancers.

In November, 2016, the Food and Drug Administration (FDA) approved nivolumab for the treatment of participants with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN). Lirilumab is not FDA approved as of now.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically or cytologically confirmed locoregionally recurrent squamous cell carcinoma of the head and neck (including any primary site, such as oral cavity, oropharynx, larynx or hypopharynx, and nasopharyngeal carcinoma)
* Must be a candidate for salvage surgery
* Willing to provide blood and tissue from diagnostic biopsy and at the time of surgery
* Has documented disease-free interval (DFI) > 8 weeks after completion of initial therapy; DFI is from the time of completion of initial treatment to the diagnosis of local or locoregional recurrence
* Any HPV status or smoking history is permitted. Oropharyngeal cancer patients are required to undergo HPV testing with p16 immunohistochemistry and/or confirmatory HPV PCR or ISH testing
* Age 18 years or older
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participant must have normal organ and marrow function as defined below within 21 days prior to study registration:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤2.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception. WOCBP should plan to use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 iu/l or equivalent units of hcg) within 24 hours prior to the start of nivolumab
* "Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

Exclusion Criteria:

* Existing significant autoimmune conditions. Patients with a history of Hashimoto thyroiditis who are stable on replacement hormone therapy are not excluded. Patients cannot be on long-term (> 4 weeks) corticosteroids at doses exceeding prednisone 20 mg (or its equivalent) prior to enrollment. Short-term corticosteroid dosing is permitted as long as steroids are discontinued within 2 weeks of study enrollment.
* Subject who has had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Subject who has been treated with immunotherapy. This includes prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Subject with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, baseline brain imaging is not required prior to enrollment in the study if patients are asymptomatic.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known human immunodeficiency virus carrier or a diagnosis of immunodeficiency. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, eg, Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
* Known non-infectious pneumonitis or any history of interstitial lung disease.
* Receipt of a live vaccine within 30 days of start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2026-07-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period March 2018 to May 2020
Groups:
- Nivolumab+Lirilumab: * The drugs will be administered intravenously. A single dose of Nivolumab and Lirilumab will be administered prior Salvage surgical resection.
  * In Cycle 1-3: Nivolumab will be administered on Days 1 and 15 and lirilumab will be administered on Day 1 of each 28 day long cycle
  * In Cycle 4-6 and beyond: Nivolumab and lirilumab will be administered on Day 1 of each 28 day long cycle.
  Nivolumab: Nivolumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells
  Lirilumab: Lirilumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells
Period: Overall Study
Arm/Group | Nivolumab+Lirilumab
Started | 29
Treated | 28
Completed | 18
Not Completed | 11
Not completed — Ineligible | 1
Not completed — Disease Progression | 2
Not completed — Withdrew Consent | 4
Not completed — Non-Compliance | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 66 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: 1-Year Disease-Free Survival Percentage
Description: The percentage of patients who were alive and disease free at one year past salvage surgery. Patients who were alive at last contact prior to the one year mark are censored. Data analysis conducted through Kaplan Meier methods.
Time Frame: 1 year since salvage surgery, up to 1 year and 23 days since treatment start
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
percentage of participants | 55.2 [34.8 to 71.7]

2. Secondary Outcome: Response at Time of Salvage Surgery
Description: Response is classified using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
  Complete Response - Disappearance of all lesions and pathologic lymph nodes.
  Partial Response - At least 30% decrease in sum of longest diameters (SLD) for the target lesions, no new lesions, and no progression of non-target lesions.
  Progressive Disease - At least 20% increase in SLD compared to smallest SLD in study or progression of non-target lesions or development of new lesions
  Stable Disease - No Partial Response and no Progressive Disease.
Time Frame: At the time of salvage surgery, up to 23 days from treatment start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
Participants
  Stable Disease | 27
  Progressive Disease | 1

3. Secondary Outcome: Median Disease-Free Survival Rate
Description: The median time that patients were alive and disease free after salvage surgery. Patients who were alive at last contact are censored at last contact. Data analysis conducted through Kaplan Meier methods
Time Frame: Up to 27.2 months post salvage surgery, up to 28 months total.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
months | 12.9 [8.18 to NA] — The last patient was censored at 27.2 months and therefore an upper limit was not reached due to an insufficient number of participants with events at data cutoff.

4. Secondary Outcome: 1-Year Overall Survival Percentage
Description: Percentage of participants who were alive at 1 year since salvage surgery. Patients alive at last contact prior to 1 year were censored.
Time Frame: 1 year post salvage surgery, up to 1 year and 23 days post treatment start.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
percentage of participants | 85.7 [66.3 to 94.4]

5. Secondary Outcome: Median Change in Programmed Cell Death Ligand - 1 Combined Positive Score
Description: The median change in Programmed Cell Death Ligand - 1 Combined Positive Score (PD-L1 CPS) from baseline to surgery. The score is derived from tumor tissue samples that measures the presence of both tumor and immune cell staining for the PD-L1 marker. Scored from 0-100, a higher score suggests the patient might respond better to treatment. A pathological responder is defined as having less than 50% viable tumor at the time of surgery.
Time Frame: Measured at baseline and then at time of salvage surgery, up to 23 days.
Population: Outcomes were compared among responders and non-responders.
Measure: Median (Full Range); unit: score
Arm/Group | Nivolumab+Lirilumab
Number analyzed (Participants) | 28
score
  Responder: number analyzed (Participants) | 12
  Responder | 2.5 [-45 to 75]
  Non-Responder: number analyzed (Participants) | 16
  Non-Responder | 0 [-45 to 49]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored for 1 year post salvage surgery, up to 1 year and 23 days post treatment start. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored from baseline to end of adjuvant therapy, up to 9 months.
Description: A serious adverse event is classified using physician's discretion. All adverse events resulting in death, life threatening events, significant disability, prolonged hospitalization, congenital abnormality/birth defect, or new cancer will be considered a serious adverse event.
Arm/Group | Nivolumab+Lirilumab
All-Cause Mortality (participants affected / at risk) | 7/28
Serious Adverse Events (participants affected / at risk) | 12/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Lirilumab (N=28)
Cardiac arrest (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Infusion related reaction (General disorders) | 1
Lung infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Lirilumab (N=28)
Anemia (Blood and lymphatic system disorders) | 7
Sinus bradycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 8
Hearing impaired (Ear and labyrinth disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 18
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 27
Esophageal stenosis (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral cavity fistula (Gastrointestinal disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 9
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Chills (General disorders) | 6
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 20
Fever (General disorders) | 5
Gait disturbance (General disorders) | 3
Infusion related reaction (General disorders) | 2
Localized edema (General disorders) | 2
Neck edema (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 14
General disorders and administration site conditions - Other, specify (General disorders) | 1
Biliary tract infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Mucosal infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 3
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 3
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 4
Weight loss (Investigations) | 3
Investigations - Other, specify (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 10
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphonia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Movements involuntary (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Presyncope (Nervous system disorders) | 2
Vasovagal reaction (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 15
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03341936/Prot_SAP_000.pdf